CLINICAL TRIAL: NCT05685641
Title: Implementation Protocol for Rapid Diagnostic Tests for Opportunistic Infections in Reference Centers in Mexico City
Brief Title: Point of Care Tests to Identify Opportunistic Infections in Advanced HIV Patients in Mexico City
Acronym: PREVALIOCDMX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Collaborators: National Institute of Cancerology (Other Government); Hospital General Dr. Manuel Gea González (Other Government); National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 181250
Record Dates: First submitted 2022-12-21; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Acquired Immunodeficiency Syndrome; Histoplasmosis AIDS; Tuberculosis Infection; Cryptococcal Meningitis
Keywords: Rapid Diagnostic Tests; Point-of-Care Systems
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Latent Tuberculosis; Meningitis, Cryptococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention group (Experimental): All enrolled patients will be included in this arm of the study, patients will be administered all rapid diagnostic tests as part of their diagnostic work-up (this will constitute the main intervention of the study)
  Interventions: Diagnostic Test: Histoplasma Urine Antigen Lateral Flow Antigen test; Diagnostic Test: Cryptococcal Lateral Flow Antigen test; Diagnostic Test: Tuberculosis-lipoarabinomannan Lateral Flow Antigen test

INTERVENTIONS:
Diagnostic Test: Histoplasma Urine Antigen Lateral Flow Antigen test — Lateral Flow Antigen test for urine samples to detect Histoplasma capsulatum disseminated disease
Diagnostic Test: Cryptococcal Lateral Flow Antigen test — Lateral Flow Antigen test for serum or cerebrospinal fluid samples to detect Cryptococcus sp meningitis or disseminated disease
Diagnostic Test: Tuberculosis-lipoarabinomannan Lateral Flow Antigen test — Lateral Flow Antigen test for serum samples to detect Mycobacterium tuberculosus disease

SUMMARY:
In Mexico City, the main cause of mortality among people living with HIV (PLHIV) continues to be opportunistic infections (OIs). Early detection of OIs allows their timely treatment and improves their prognosis. The use of rapid diagnostic tests (RDT) based on antigens of the most frequent causative agents of OIs allows adequate screening of these patients and facilitates decision making at the point of care. Unfortunately, these studies are not widely available in the different PLHIV care centers in the CDMX. We will conduct an open-label, non-inferiority uncontrolled clinical trial to investigate the diagnostic performance of urinary lipoarabinomannan, urinary Histoplasma antigen and serum Cryptococcus antigen in patients presenting for care with advanced HIV in CDMX, supported by rapid cluster of differentiation 4 (CD4) testing with lateral flow technology. Four referral hospitals will participate over 12 months. All patients with diagnosed HIV disease and suspected advanced disease presenting for care at participating centers will be included in the study. An inventory of approximately 1000 RDT will be obtained and distributed among the participating sites. A study coordinator will be hired and will visit each site once a week to collect the study variables and follow up on the included patients. The primary outcome of the study will be the percentage of patients with advanced disease who present with diagnoses made by RDT compared to historical controls of patients diagnosed with OI in 2022 at participating centers by conventional methods. Secondary outcomes will be time to initiation of antiretroviral therapy (ART), time to initiation of OI treatment, and 30-day mortality after HIV diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Positive ELISA test or positive viral load for HIV.
* Patients with suspected or confirmed advanced HIV disease defined as follows:

  * Confirmed: asymptomatic patients with CD4 count less than 200 cells/ml within 3 months of study inclusion or confirmed diagnosis of an AIDS-defining opportunistic illness within the last 3 months.
  * Suspected: patients who, irrespective of CD4 count, present any symptoms suggestive of systemic infection that, at the discretion of the treating physicians, produce suspicion of an AIDS-defining opportunistic disease (e.g., fever, productive cough, diaphragmatic diapers, etc.). Fever, productive cough, nocturnal diaphoresis, altered mental status, headache, lymphadenopathy, dermatological lesions) or that meet criteria for HIV wasting syndrome (loss of 10% of baseline weight plus the presence of chronic diarrhea or chronic weakness and an episode of fever in the last 30 days).
* Patients without effective antiretroviral therapy defined as not having received antiretroviral treatment in the last 3 months or in virologic failure (2 consecutive viral loads with more than 1000 copies/ml).

Exclusion Criteria:

* Patients with a viral load of less than 1000 copies/ml.
* Patients presenting for care having started treatment for systemic mycoses (amphotericin B or azoles) and tuberculosis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Time until opportunistic infection treatment initiation | 30 days
  Amount of time in days from the diagnosis of the opportunistic infection until the initiation of the specific treatment for the detected infection

SECONDARY OUTCOMES:
AIDS-related mortality at 30 days | 30 days
  If a patient has died due to AIDS-related causes
AIDS-related mortality at 90 days | 90 days
  If a patient has died due to AIDS-related causes
Monthly incidence of histoplasmosis, cryptococcosis and tuberculosis | Through study completion, an average of 1 year
  The amount of diagnosed cases of histoplasmosis, cryptococcosis and tuberculosis per amount of advanced HIV-patients seen every month in the study sites
Time until antiretroviral treatment initiation | 30 days
  Days passed from a patient's HIV diagnosis until he is given antiretroviral treatment for the first time

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Camiro Zúñiga, MD, Principal Investigator — Centro Medico ABC
Locations (4):
- Mexico (4):
  - General Hospital Dr. Manuel Gea Gonzalez, Mexico City
  - National Center of Nutrition and Medical Sciences, Mexico City
  - National Institute of Cancerology, Mexico City
  - National Institute of Respiratory Diseases, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be uploaded to a public database sharing website
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made publicly available after publishing of the study in a peer reviewed journal
Access Criteria: Data will be made available upon request